CLINICAL TRIAL: NCT02613338
Title: Kinematic Analysis: Posterior Stabilized, Fixed Bearing Total Knee Arthroplasty With Attune Knee System - Phase 2
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Fred M. Roddy Professor of Biomedical Engineering, The University of Tennessee, Knoxville
Other Study IDs: 9568FB; IIS-13002 (Other Grant/Funding Number: DePuy Synthes)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DePuy Attune PS FB knee system: Patients implanted with a DePuy Attune posterior stabilizing fixed bearing knee system
  Interventions: Device: DePuy Attune posterior stabilizing fixed bearing knee system

INTERVENTIONS:
Device: DePuy Attune posterior stabilizing fixed bearing knee system — Individuals implanted with the DePuy Attune posterior stabilizing fixed bearing knee system at least three months post-operative.

SUMMARY:
A better understanding of knee joint kinematics is important to explain the premature polyethylene wear failures within total knee arthroplasties (TKAs) and to help design a prosthesis that most closely approximates the normal knee. Specifically, posterior stabilizing (PS) knees have been found to be associated with lower amounts of posterior femoral rollback, higher occurrence of reverse axial rotation and increased amount of condylar lift-off. The DePuy Synthes Joint Reconstruction's Attune PS fixed bearing (FB) knee system has incorporated subtle changes in its design to address restoration of kinematics that more closely resemble those of a normal knee. To understand if this design is able to effectively restore kinematics in the implanted knee, further in vivo analysis is necessary. This continuation of the study will analyze 30 subjects with the Attune PS FB 3 months post-operatively using the University of Tennessee's mobile fluoroscopy unit while performing three daily activities, level walking, ramp down and deep knee bend.

ELIGIBILITY:
Inclusion Criteria:

* At least three (3) months post-operative with no other surgical procedures conducted within the past six months

  * Between 30-80 years of age
  * Body weight of less than 280 lbs
  * Must be between 160cm (5'3) and 193cm (6'4) tall
  * Body Mass Index (BMI) >18.5 and <35
  * Judged clinically successful with a Knee Society score (KSS) of greater than 80
  * Have good-to-excellent post-operative passive flexion with no ligamentous laxity or pain
  * Must be able to walk on level ground without aid of any kind, perform a ramp descent, and a deep knee bend (DKB), all without assistance
  * Will have a DePuy Attune PS TKA

Exclusion Criteria:

* Pregnant or potentially pregnant females will be excluded from the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals implanted with the DePuy Attune posterior stabilizing fixed bearing knee system at least three months post-operative.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrija Sharma, Ph. D., Principal Investigator — University of Tennessee; William R Hamel, Ph. D., Principal Investigator — University of Tennessee
Locations (5):
- United States (5):
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Abercrombie Radiology, Knoxville, Tennessee
  - Dougherty Engineering Building, Room M007, Knoxville, Tennessee
  - Perkins Hall, The University of Tennessee, Knoxville, Tennessee
  - Science and Engineering Research Facility, The University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DePuy Attune PS FB Knee System
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.48 (5.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Femoro-tibial Kinematics - Lateral Anterior/Posterior Motion
Description: Amount of anterior sliding (positive) and/or posterior rollback (negative) of the lateral condyle during DKB, gait, and ramp down
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
mm
  Deep Knee Bend | -5.81 (3.12)
  Gait | -0.1 (1.57)
  Ramp Down | 0.58 (1.71)

2. Primary Outcome: Femoro-tibial Kinematics - Medial Anterior/Posterior Motion
Description: Amount of anterior sliding (positive) and/or posterior rollback (negative) of the medial condyle during DKB, gait, and ramp down
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
mm
  Deep Knee Bend | -1.81 (2.04)
  Gait | -0.07 (1.82)
  Ramp Down | -0.14 (1.39)

3. Secondary Outcome: Max Ground Reaction Force - Deep Knee Bend
Description: Collected simultaneously with fluoroscopy data, ground reaction forces were obtained using a force plate (fixed to the ground) while subject performed activity. Maximum force measured in the vertical direction measured during the activity was normalized with respect to participant's body weight and has been termed "maximum reaction force."
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: proportion of body weight
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
proportion of body weight | 0.83 (0.17)

4. Secondary Outcome: Max Ground Reaction Force - Gait
Description: Collected simultaneously with fluoroscopy data, ground reaction forces were obtained using a force plate (fixed to the ground) while subject performed activity. Maximum force measured in the vertical direction measured during the activity.
  was normalized with respect to participant's body weight and has been termed "maximum reaction force."
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: proportion of body weight
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
proportion of body weight | 1.09 (0.23)

5. Secondary Outcome: Max Ground Reaction Force - Ramp Down
Description: as for outcome 4
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: proportion of body weight
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
proportion of body weight | 1.06 (0.21)

6. Primary Outcome: Femoro-tibial Kinematics - Axial Rotation
Description: Amount of axial rotation of the femoral component with respect to the tibial component during DKB, gait, and ramp down. Positive indicated external rotation of femur wrt tibia.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
degrees
  Deep Knee Bend | 5.4 (4.04)
  Gait | 0.17 (2.46)
  Ramp Down | 0.88 (4.36)

7. Primary Outcome: Femoro-tibial Kinematics - Weight-bearing Flexion
Description: Amount of weight-bearing flexion during DKB, gait, and ramp down. All numbers are positive, indicating magnitude.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DePuy Attune PS FB Knee System
Number analyzed (Participants) | 30
degrees
  Deep Knee Bend | 110.27 (20.40)
  Gait | 28.5 (9.85)
  Ramp Down | 33.8 (8.38)

ADVERSE EVENTS:
Time Frame: 3 years, one month
Arm/Group | DePuy Attune PS FB Knee System
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02613338/Prot_SAP_000.pdf